CLINICAL TRIAL: NCT05180227
Title: Targeted Transcutaneous Stimulation to Restore Autonomic Cardiovascular Health in Veterans With Spinal Cord Injury
Brief Title: Transcutaneous Stimulation in Spinal Cord Injury
Acronym: SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: B3706-M; IK1RX003706 (NIH)
Record Dates: First submitted 2021-11-19; First posted 2022-01-06 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury
Keywords: Blood pressure; Orthostatic hypotension; Transcutaneous stimulation; Cardiovascular disease
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension, Orthostatic; Cardiovascular Diseases | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: All participants will complete transcutaneous stimulation mapping sessions to determine the optimal parameters to increase and maintain systolic blood pressure between 110-130 mmHg.
Who Masked: Participant
Masking Description: Participants will be blinded to which stimulation parameters they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Without Stimulation (No Intervention): Seated blood pressure without transcutaneous spinal cord stimulation will be assessed.
- With Stimulation (Active Comparator): Seated blood pressure with transcutaneous spinal cord stimulation will be assessed.
  Interventions: Device: DS8R

INTERVENTIONS:
Device: DS8R — transcutaneous stimulation of the spinal cord.
  Other Names: Transcutaneous Stimulation
  Arms: With Stimulation

SUMMARY:
Cardiovascular disease has become the leading cause of death in the spinal cord injury population. Increased reliance on the renin-angiotensin-aldosterone system (RAAS) is believed to decrease falls in blood pressure when moving from a laying down position to upright; however, findings in the general population link the RAAS with remodeling and restructuring of the arterial walls. Therefore, intervention to stabilize and normalize blood pressure should be a priority in individuals with spinal cord injury who have low blood pressure. Advances in stimulation on the skin of the spinal cord offer an approach to restore cardiovascular control and improve blood pressure regulation; however, electrode placement and stimulation parameters needed to increase blood pressure are not well understood. Therefore, the aim of the study is to identify placement of electrodes on the skin, and frequency and amplitude of the stimulation to regulate blood pressure.

DETAILED DESCRIPTION:
Although life expectancies have improved in the SCI population, longevity remains below the general population, due to increased incidence of cardiovascular disease, which is the leading cause of mortality in individuals with chronic SCI. Autonomic nervous system dysfunction and blood pressure instability contribute to the increased cardiovascular disease risk in the SCI population; however, because a majority of individuals with SCI remain asymptomatic the diagnosis and treatment of blood pressure instability is not a clinical priority. This is due, in part, to lack of safe and effective interventions, even though mounting evidence strongly supports adverse effects of blood pressure instability on the cerebral circulation, cognitive function, and quality of life. Identifying individualized transcutaneous stimulation parameters that safely and effectively increase and stabilize blood pressure in hypotensive individuals with SCI will provide the foundational evidence to support eventual wide-spread clinical utility throughout the VA healthcare system. 10 participants who are cleared, will go through multiple mapping sessions to find out the most appropriate electrode placement to increase seated blood pressure. The study will take approximately 1 to 13 study visits, of between 3-5 hours, per participant.

ELIGIBILITY:
Inclusion Criteria:

* above the age of 18 years old
* individuals with traumatic spinal cord injuries at or above T6

  * duration of injury if more than 1 year
  * non-ambulatory
  * American spinal injury association scale A, B or C
* able to provide consent
* non-ventilator
* hypotensive (males: systolic blood pressure less than 110 mmHg and/or diastolic blood pressure less than 70 mmHg; females: systolic blood pressure less than 100 mmHg and/or diastolic blood pressure less than 70 mmHg)

Exclusion Criteria:

* acute illness or infection
* documented history of controlled or uncontrolled diabetes
* any other neurological disease other than spinal cord injury
* cardiovascular disease (coronary artery disease, congestive heart failure, peripheral artery disease, stroke)
* present of history of thrombosis in the last 12 months, severe contractures
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caitlyn Peters, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peters CG, Harel NY, Weir JP, Wu YK, Murray LM, Chavez J, Fox FE, Cardozo CP, Wecht JM. Transcutaneous Spinal Cord Stimulation to Stabilize Seated Systolic Blood Pressure in Persons With Chronic Spinal Cord Injury: Protocol Development. Neurotrauma Rep. 2023 Dec 19;4(1):838-847. doi: 10.1089/neur.2023.0063. eCollection 2023. PMID 38156073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 potential participants were screened and enrolled between June 2022 and December 2023.
Groups:
- People With Spinal Cord Injury: People with chronic spinal cord injury undergoing spinal cord stimulation to increase and stabilize seated systolic blood pressure.
Period: Overall Study
Arm/Group | People With Spinal Cord Injury
Started | 10
Completed | 8
Not Completed | 2
Not completed — Hypertension at screening | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants Receiving Spinal Cord Stimulation to Increase and Stabilize Systolic Blood Pressure: Demographic, ethnic and spinal cord injury-specific characteristics of the participants enrolled in the trial
Arm/Group | Participants Receiving Spinal Cord Stimulation to Increase and Stabilize Systolic Blood Pressure
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Neurological level of spinal cord injury [Count of Participants; unit: Participants] — This was determined using the International Standards for Neurological Classification of Spinal Cord Injury exam (Kirshblum et al., 2011).
  Participants
    Cervical | 7
    Thoracic | 3
AIS classification of injury [Count of Participants; unit: Participants] — American Spinal Injury Association Impairment Scale (AIS) classification is determined with the International Standards for Neurological Classification of Spinal Cord Injury exam (Kirshblum et al., 2011). AIS A - no sensory or motor function below the neurological level of spinal cord injury; AIS B - sensory, but no motor function preserved below the neurological level of spinal cord injury; AIS C - sensory and partial motor function preserved below the neurological level of spinal cord injury.
  Participants
    AIS A | 4
    AIS B | 4
    AIS C | 2
Time since injury [Mean (Standard Deviation); unit: years] | 15.9 (16.8)

OUTCOME MEASURES:

1. Primary Outcome: Seated Systolic Blood Pressure
Description: Seated systolic blood pressure response to spinal cord stimulation at T7/T8, T9/10, T11/12, L1/L2) to determine the best cathode electrode placement on the spine that increases systolic blood pressure between 110-130 mmHg.
Time Frame: From enrollment to the end of the last study visit, approximately 30 days.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- No Stimulation: Seated blood pressure will be assessed without TSCS.
- T7/8: Seated blood pressure assessed with TSCS at T7/8.
- T9/10: Seated blood pressure assessed with TSCS at T9/10.
- T11/12: Seated blood pressure assessed with TSCS at T11/12.
- L1/2: Seated blood pressure assessed with TSCS at L1/2.
Arm/Group | No Stimulation | T7/8 | T9/10 | T11/12 | L1/2
Number analyzed (Participants) | 8 | 8 | 6 | 6 | 6
mmHg | 86 (16.6) | 100.4 (13.9) | 102.7 (13.2) | 101.3 (11.8) | 102.1 (13.5)

ADVERSE EVENTS:
Time Frame: From enrollment until end of last study visit, up to 30 days.
Groups:
- Stimulation: Participant will have seated blood pressure monitored without and with transcutaneous stimulation.
  DS8R: transcutaneous stimulation of the spinal cord.
Arm/Group | Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stimulation (N=10)
Superficial skin burn (Skin and subcutaneous tissue disorders) | 3 (9) — Superficial redness and irritation of the skin under the stimulating electrode.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT05180227/Prot_001.pdf
  • Statistical Analysis Plan (2025-08-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT05180227/SAP_002.pdf
  • Informed Consent Form (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT05180227/ICF_000.pdf